CLINICAL TRIAL: NCT02551770
Title: Straumann® Emdogain® Application In Conjunction With Minimally Invasive Surgical Technique For Periodontal Disease Treatment: A Split-Mouth Design Study
Brief Title: Emdogain Minimally Invasive Surgical Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Straumann AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR 01/15
Record Dates: First submitted 2015-09-14; First posted 2015-09-16 (Estimated); Results first posted 2019-10-17 (Actual); Last update posted 2019-10-17 (Actual); Status verified 2019-10

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis | interventions — Tooth Exfoliation; Root Planing; enamel matrix proteins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test (with Emdogain) (Active Comparator): Scaling and root planing with Emdogain
  Interventions: Procedure: Scaling and root planing; Device: Emdogain application
- Control (without Emdogain) (Other): Scaling and root planing without Emdogain
  Interventions: Procedure: Scaling and root planing without Emdogain

INTERVENTIONS:
Procedure: Scaling and root planing — Using minimally invasive surgical procedure (scaling and root planing) with Emdogain application to treat one contra-lateral quadrant in subject's jaw.
  Arms: Test (with Emdogain)
Procedure: Scaling and root planing without Emdogain — Using minimally invasive surgical procedure (scaling and root planing) without Emdogain application to treat one contra-lateral quadrant in subject's jaw.
  Arms: Control (without Emdogain)
Device: Emdogain application — Using minimally invasive surgical procedure (scaling and root planing) with Emdogain application to treat one contra-lateral quadrant in subject's jaw
  Arms: Test (with Emdogain)

SUMMARY:
The aim of this controlled study is to assess the clinical outcomes and patient reported outcomes of using minimally invasive surgical procedure with Straumann Emdogain as an adjunct (test treatment) or without Straumann Emdogain (control treatment).

DETAILED DESCRIPTION:
The aim of the study will be achieved through the following primary and secondary objectives. The primary objective is to evaluate the regenerative potential of Straumann Emdogain by comparing the change in clinical attachment level from baseline to 12 months between the test and control arms. The regenerative potential of Straumann Emdogain will also be assessed by comparing the changes in gingival margins, changes in average probing pocket depth, changes in full mouth plaque score, changes in bleeding on probing, and changes in root dentin hypersensitivity from baseline to 12 months between the test and control arms.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have voluntarily signed the informed consent form before any study related procedures
* Subjects must be males or females who are 18-85 years of age
* Subjects must have moderate to severe chronic, generalized periodontitis with pockets of 5 mm - 8mm probing depth in at least 2 pockets per contralateral quadrants in one arch (study teeth)
* Subjects must be committed to the study and the required follow-up visits
* Subjects must be in good general health as assessed by the Investigator

Exclusion Criteria:

* Subjects taking or intending to take any medications during the duration of the study that will potentially affect healing and inflammation
* Subjects who are currently heavy smokers (defined >10 cigarettes per day or >1 cigar per day) or who use chewing tobacco
* Subjects being treated with systemic antibiotics or subjects that were treated with systemic antibiotics within 3 months prior to treatment in this study
* Subjects with uncontrolled diabetes
* Subjects that are immunocompromised or immunosuppressed
* Subjects that cannot provide informed consent
* Subjects with drug or alcohol abuse
* Subjects that have undergone periodontal root planing or periodontal surgery in the last 6 months
* Subjects that are pregnant
* Subjects with necrotizing periodontitis or periodontitis related to systemic disease
* Teeth with pockets with probing depth ≥ 9 mm will not classify as study teeth
* Teeth with pockets or defects with furcation involvement will not classify as study teeth
* Teeth with mobility degree > 1 without splint will not classify as study teeth
* Subjects with test and control sites in the two quadrants on adjacent teeth
* Patients with compromised health conditions such as diabetes, systemic diseases, high dose steroid therapy, bone metabolic diseases, radiation or immune-oppressive therapy, and infections or vascular impairment at the surgical site
* Subjects with conditions or circumstances, in the opinion of the Investigator , which would prevent completion of study participation or interfere with analysis of study results

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2019-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela K McClain, DDS, Principal Investigator — Periodontics and Implant Dentistry; Veronique Benhamou, DDS, Principal Investigator — Clinique Paro Excellence; Jennifer H Doobrow, DMD, Principal Investigator — Periodontal & Implant Associates
Locations (4):
- United States (2):
  - Periodontal and Implant Associates, Inc., Cullman, Alabama
  - Periodontics and Implant Dentistry, Aurora, Colorado
- Clinique Paro Excellence, Montreal, Quebec, Canada
- Universitätsmedizin der Johannes Gutenberg Universität Mainz, Mainz, Germany

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Oversight. 1 extra patient was enrolled.
Units Other Than Participants: Study Teeth
Period: Overall Study
Arm/Group | Test (With Emdogain) | Control (Without Emdogain)
Started | 51; 167 Study Teeth | 51; 170 Study Teeth
Completed | 48; 162 Study Teeth | 48; 162 Study Teeth
Not Completed | 3; 5 Study Teeth | 3; 8 Study Teeth

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Participants assigned to receive both interventions (i.e., control and test) in different quadrants of the jaw.
  - Test Treatment (Scaling and root planing with Emdogain): Scaling and root planing: Using minimally invasive surgical procedure (scaling and root planing) with Emdogain application to treat one contra-lateral quadrant in subject's jaw.
  Emdogain application: Using minimally invasive surgical procedure (scaling and root planing) with Emdogain application to treat one contra-lateral quadrant in subject's jaw.
  - Control Treatment (Scaling and root planing): Scaling and root planing: Using minimally invasive surgical procedure (scaling and root planing) to treat one contra-lateral quadrant in subject's jaw.
Arm/Group | All Participants
Number analyzed (Participants) | 51
Age, Customized [Number; unit: Participants]
  <18 | 0
  18-85 | 51
  >85 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 50
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 45
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Canada | 4
  United States | 32
  Germany | 15

OUTCOME MEASURES:

1. Primary Outcome: Change in Clinical Attachment Levels (CAL)
Description: CAL will be measured in millimeters on the study teeth at 6 locations. Outcome is mean change of CAL from baseline measurements at surgery to 12-months post-surgery, taken from the deepest pocket of a patient's test and control teeth measured at baseline. Analysis will compare the mean change of CAL for test and control treatment arms.
Time Frame: Baseline and 12 Month Follow-Up Visit
Population: The ITT data set with imputation of missing values (five CAL values were missing at 12 month follow-up and were replaced with values from 9 month follow-up).
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Test (With Emdogain) | Control (Without Emdogain)
Number analyzed (Participants) | 49 | 49
mm | -2.2 (1.5) | -2.1 (1.3)

2. Secondary Outcome: Change in Gingival Margin (GM)
Description: GM will be measured in millimeters on the study teeth at 6 locations. Outcome is mean change of GM from baseline at surgery to 12-months-post surgery, taken from the deepest pocket of a patient's test and control teeth measured at baseline. Analysis will compare the mean change of GM for test and control treatment arms.
Time Frame: Baseline and 12 Month Follow-Up Visit
Population: from the ITT dataset. Missing data was not entered.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Test (With Emdogain) | Control (Without Emdogain)
Number analyzed (Participants) | 47 | 46
mm | -.3 (.9) | -.2 (1.0)

3. Secondary Outcome: Change in Pocket Probing Depth (PPD)
Description: PPD will be measured in millimeters on the study teeth in 6 locations. Outcome is mean change of PPD from baseline at surgery to 12-months post-surgery, taken from the deepest pocket of a patient's test and control teeth at baseline. Analysis will compare the mean change of PPD for test and control treatment arms.
Time Frame: Baseline and 12 Month Follow-Up Visit
Population: ITT dataset.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Test (With Emdogain) | Control (Without Emdogain)
Number analyzed (Participants) | 47 | 47
mm | -2.4 (1.3) | -2.3 (1.2)

4. Secondary Outcome: Change in Full Mouth Plaque Score (FMPS)
Description: FMPS will be calculated based on the number of tooth surfaces with plaque over the total number of tooth surfaces x 100. The value is presented as a percent. The difference in FMPS between 12 months and baseline will be determined.
Time Frame: Baseline and 12 Month Follow-Up Visit
Population: ITT data set.
Measure: Number; unit: Full Mouth Plaque Score
Units Other Than Participants: Tooth surfaces
Arm/Group | Test (With Emdogain) | Control (Without Emdogain)
Number analyzed (Participants) | 51 | 51
Number analyzed (Tooth surfaces) | 668 | 684
Full Mouth Plaque Score
  Baseline | 54.34 | 55.17
  12 Month Follow Up: number analyzed (Tooth surfaces) | 612 | 604
  12 Month Follow Up | 35.03 | 31.58

5. Secondary Outcome: Change in Bleeding on Probing (BoP)
Description: For the categorical variable BoP, the frequency of bleeding (present or absent) will be counted (absolute and in percent) over all measured sites around the identified study teeth for each treatment group. The results will be compared between the 12-month follow-up and baseline.
Time Frame: Baseline and 12 Month Follow-Up Visit
Population: ITT data set.
Measure: Count of Units; unit: Sites
Units Other Than Participants: Sites
Arm/Group | Test (With Emdogain) | Control (Without Emdogain)
Number analyzed (Participants) | 51 | 51
Number analyzed (Sites) | 1002 | 1026
Sites
  Baseline sites with bleeding | 547 | 576
  Baseline sites without bleeding | 455 | 450
  12 month sites with bleeding: number analyzed (Sites) | 969 | 966
  12 month sites with bleeding | 172 | 223
  12 month sites without bleeding: number analyzed (Sites) | 969 | 966
  12 month sites without bleeding | 797 | 743

6. Secondary Outcome: Change in Root Dentin Hypersensitivity
Description: Presence of root dentin hypersensitivity will be recorded as "none" (no reaction from the subject), "mild" (sensible with no pain), "moderate" (sensible with slight pain), or "severe" (sensible with pain that persists for a while) after a conventional air blast is applied to the study tooth. Changes in the frequency of categories will be determined and compared between the two treatment arms. An improvement is defined as a decreased reaction (for example, severe to mild), a deterioration is defined as increased reaction (for example, none to moderate), and unchanged is no change to reaction (for example, mild to mild).
Time Frame: Baseline and 12 Month Follow-Up Visit
Population: ITT data set study teeth. Baseline collected at either visit 1 or visit 2 based on different versions of CIP.
Measure: Count of Units; unit: Study Teeth
Units Other Than Participants: Study Teeth
Arm/Group | Test (With Emdogain) | Control (Without Emdogain)
Number analyzed (Participants) | 51 | 51
Number analyzed (Study Teeth) | 159 | 156
Study Teeth
  Improvement in Root Dentin Hypersensitivity | 44 | 37
  Deterioration in Root Dentin Hypersensitivity | 8 | 13
  Unchanged Root Dentin Hypersensitivity | 107 | 106

7. Secondary Outcome: Change in Post-surgical Pain
Description: Post-surgical pain will be measured on a 100 millimeter visual analog scale. The range is 0 (no pain) to 99 (nearly maximum pain). The lower the value, the better the outcome. The subjects will be instructed to mark their level of pain on a line for both the test quadrant and the control quadrant. The average change in pain level will be determined and compared between the two arms.
Time Frame: 1-2 days post surgery, 1 week post surgery, and 2 weeks post surgery
Population: ITT dataset.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Test (With Emdogain) | Control (Without Emdogain)
Number analyzed (Participants) | 49 | 49
mm
  Pain Level 1-2 days post sx. | 14.3 (22.6) | 12.9 (20.9)
  Pain level 1 week post sx | 9.8 (20.6) | 8.1 (19.6)
  Pain Level 2 weeks post sx. | 6.0 (16.6) | 5.0 (13.8)

ADVERSE EVENTS:
Time Frame: Up to 12 months.
Description: All participants received both interventions and adverse events were not collected with regard to separate intervention.
Groups:
- All Participants: All Participants
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/51
Serious Adverse Events (participants affected / at risk) | 1/51
Other Adverse Events (participants affected / at risk) | 15/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=51)
Breast Cancer diagnosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Subject diagnosed with breast cancer. Unrelated to device or procedure
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=51)
Sinus Infection (Infections and infestations) | 2 (2) — Subject reported sinus infection. Unrelated to device or procedure.
Extensive tooth decay (General disorders) | 1 (1) — Extensive tooth decay site #31. Unrelated to device or procedure.
Cold/Flu (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Cold/Flu. Unrelated to device or procedure.
Mild discomfort when chewing (General disorders) | 1 (1) — mild discomfort with chewing. Possibly related to procedure.
Retrained bony sequestrum (General disorders) | 1 (1) — Retained bony sequestrum. Unrelated to device or procedure.
Generalized sensation of burning mouth (General disorders) | 1 (1) — Generalized sensation of burning mouth. Unrelated to device or procedure.
Itching skin reaction gum (General disorders) | 1 (1) — Itching skin reaction gum. Possibly related to device or procedure.
Itching skin reaction neck area, external (Skin and subcutaneous tissue disorders) | 1 (1) — Itching skin reaction neck area, external, no pain. Possibly related to device.
Fracture of Veneer #21 (General disorders) | 1 (1) — Fracture of veneer #21. Unrelated to device or procedure.
Hematoma (General disorders) | 1 (1) — Hematoma right side above tooth # 5 and #6. Approx 2-3 cms big. No pain. Definitely related to procedure.
Tooth fracture #23 (General disorders) | 1 (1) — Tooth Fracture #23. Unrelated to device or procedure.
Apical periodontitis (General disorders) | 1 (1) — Apical periodontitis. Unrelated to device or procedure.
Abscess on extracted tooth #20 (General disorders) | 1 (1) — Abscess on tooth #20. Not study tooth. Unrelated to device or procedure.
Bleeding and mobility at #24 and 28 (General disorders) | 1 (1) — Bleeding and mobility at teeth #24 and #28. Unrelated to device or procedure.
Loosening of bridge (General disorders) | 1 (4) — Loosening of bridge. Unrelated to device or procedure.
Sensitivity to cold teeth # 4,5,7 and 9-11 (General disorders) | 1 (1) — Sensitivity to cold teeth # 4,5,7 and 9-11. Possibly related to procedure.
Unclear tooth complaint #5 and #6 (General disorders) | 1 (1) — Unclear tooth complaint #5 and #6. Unrelated to device or procedure.
Restoration prosthetic problem (General disorders) | 1 (2) — Restoration prosthetic problem. Unrelated to device or procedure.
Hypersensitivity to pain # 22 and 25-28 (General disorders) | 1 (1) — Hypersensitivity to pain #22 and 25-28. Possibly related to procedure.
Sensitivity to warmth and cold # 19,21,22,25,27-29 (General disorders) | 1 (1) — Sensitivity to warmth and cold #19,21,22,25,27-29. Definitely related to procedure.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-09): https://cdn.clinicaltrials.gov/large-docs/70/NCT02551770/Prot_SAP_000.pdf